CLINICAL TRIAL: NCT03773341
Title: Causes and Patterns of ACL Injuries Among Egyptian People
Brief Title: Causes and Patterns of Anterior Cruciate Ligament Injuries Among Egyptian Population
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali Soliman Ali, MBBCh principle investigator, Assiut University
Other Study IDs: ACL injuries
Record Dates: First submitted 2018-11-11; First posted 2018-12-12 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: ACL Injury
Keywords: ACL injury; non sport causes; Egyptians
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: research questionnaire — Patient personal data History taking clinical knee examination

SUMMARY:
The aim of work is to detect the patterns and the causes of ACL injury among Egyptian population and to identify its risk factors. Identify the male to female ratio of injuries in our community. To document the patterns and frequencies of associated injuries

DETAILED DESCRIPTION:
The ACL (Anterior Cruciate ligament) is one of the most frequently injured ligaments of the knee, with a prevalence estimated to be 1 in 3000 in the US (greater than 120000 cases annually). ACL injury frequently affects young, active individuals. It is also frequently associated with other structural injuries in the Knee joint like meniscal tears and multi-ligamentous injuries. ACL injury leads to increased laxity in the knee, predispose the knee to subsequent injuries and early onset osteoarthritis of the knee.

Sports related trauma is the commonest cause of ACL rupture. Females are reported to have 2 to 10-fold higher risk of injury than males playing the same sport. According to previous studies at Assuit University Hospital the impression was that the ACL injuries are more common in males than females. Additionally, non-sports injuries like motor cycle accidents and domestic injuries are expected to be a major cause of ACL rupture, besides sports injuries, among Egyptian population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed ACL injury

Exclusion Criteria:

* Patients with ACL injury associated with fracture at the same limb

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Egyptian patients with confirmed ACL injury by clinical and radio logical diagnoses older than 18 years old and younger than 60 years old
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Patterns of ACL injuries among Egyptian population | one year
  Detection of patterns of ACL injuries among 500 Egyptian patient older than 18 years old and younger than 60 years old e.g valgus stress, faulty landing and whether the injury is sport related or not through a validated research questionnaire

REFERENCES:
- [Background] Levine JW, Kiapour AM, Quatman CE, Wordeman SC, Goel VK, Hewett TE, Demetropoulos CK. Clinically relevant injury patterns after an anterior cruciate ligament injury provide insight into injury mechanisms. Am J Sports Med. 2013 Feb;41(2):385-95. doi: 10.1177/0363546512465167. Epub 2012 Nov 9. PMID 23144366
- [Background] Arendt E, Dick R. Knee injury patterns among men and women in collegiate basketball and soccer. NCAA data and review of literature. Am J Sports Med. 1995 Nov-Dec;23(6):694-701. doi: 10.1177/036354659502300611. PMID 8600737
- [Background] Anderson AF, Dome DC, Gautam S, Awh MH, Rennirt GW. Correlation of anthropometric measurements, strength, anterior cruciate ligament size, and intercondylar notch characteristics to sex differences in anterior cruciate ligament tear rates. Am J Sports Med. 2001 Jan-Feb;29(1):58-66. doi: 10.1177/03635465010290011501. PMID 11206258